CLINICAL TRIAL: NCT00901355
Title: Morbidity and Mortality Based on Blood Pressure and Arterial Stiffness in Institutionalized Persons Aged 80 and Over: Study PARTAGE (Predictive Values of Blood Pressure and Arterial Stiffness in Institutionalized Very Aged Population).
Brief Title: Predictive Values of Blood Pressure and Arterial Stiffness in Institutionalized Very Aged Population
Acronym: PARTAGE
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: French Cardiology Society (Other); Boehringer Ingelheim (Industry); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2006-A00042-49
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension; Elderly; Cardiovascular Mortality; Cognitive Impairment; Morbidity
Keywords: Blood pressure; Arterial stiffness; Morbidity; Mortality; Elderly
MeSH Terms: conditions — Hypertension; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Introduction: High blood pressure especially systolic hypertension is a common condition in the elderly and is considered as a major determinant not only of cardiovascular (CV) morbidity and mortality, but also of several other age-related diseases, frailty and loss of autonomy. Actually, the association between BP levels and morbidity and mortality in the very elderly persons with several co-morbidities remains a controversial issue

Objectives: The aim of the PARTAGE study (Predictive values of blood pressure and arterial stiffness in institutionalized very aged population)is to determine the predictive value of blood pressure (BP) and arterial stiffness for overall mortality, major cardiovascular events and cognitive decline in a large population of institutionalized subjects aged 80 and over.

Methods: The population is composed of 1130 subjects aged over 80, living in nursing home, included by four french university hospitals centre (Nancy, Dijon, Paris, Toulouse) and two Italian (Cesena, Verona). Subjects with severe dementia and a very low level of autonomy are excluded from the study During the first visit, blood pressure were measured using an automatic monitor by physician in sitting and standing position (clinical BP and Orthostatic BP) and by a self measurement of blood pressure 3 measurements, in the morning and the evening, during 3 consecutive days).

Arterial stiffness is evaluated by measuring the carotid-femoral and carotid-radial pulse wave velocity (PWV) with the PulsePen® automatic device. Deaths and cardiovascular events are recorded during a follow-up of 2 years.

The hypothesis of the PARTAGE longitudinal study is that in very elderly frail individuals with multiple co-morbidities, CV risk could be better evaluated by combining self-measurements of BP and direct evaluation of arterial stiffness which are less influenced by the above mentioned disease and co-morbidities.

DETAILED DESCRIPTION:
The aim of PARTAGE study (Predictive values of blood pressure and arterial stiffness in institutionalized very aged population) is to determine the predictive value of blood pressure (BP) and arterial stiffness estimated by pulse wave velocity (PWV) on overall mortality, major CV events and cognitive decline in a large population of subjects living in nursing homes aged 80 and over.

Method:

Participants are included if they are aged 80 year old and over, are institutionalized and if they have signed the informed consent.

Persons are excluded if they have severe dementia (Mini Mental Status Examination: MMSE<12), a low level of autonomy (Activity of daily living: ADL≤2) and they are under guardianship or "a measure of legal protection".

All geriatric assessment instruments and arterial measures are applied by several trained medical research teams (geriatricians, cardiologists, psychologists) present at each university hospitals centre. All medical teams received the same standard operating procedures. All the assessments are performed in the nursing homes.

Clinical data collection During the first visit in the nursing home, the medical research team collect a large amount of information during a face-to-face interview and from patient's medical records. Following information are recorded for each participant in a case report form (CRF): sociodemographic characteristics, educational level, medical history, chronic diseases (cardio vascular, central nervous system, respiratory), depressive symptoms, history of falls, co morbidity and medication use.

Additionally, a clinical examination of functional status, cognitive function, blood pressure and arterial stiffness are realized by medical research teams.

* Comorbidities are quantified using the Charlson combined comorbidity index.
* Functional status is evaluated by the Katz Index of independence in ability in activities of daily living (ADL) (bathing, dressing, going to the toilet, transferring from bed to chair, continence and feeding).
* Cognitive status was assessed using the Mini-Mental-Status-Examination (MMSE), which is a global measurement of cognitive function evaluating various dimensions of cognition (memory, calculation, orientation in space and time, language, and word recognition).

Peripheral blood pressure measurements:

Peripheral BP and heart rate (HR) are performed at brachial artery level using the validated automated oscillometric device Colson DM-H20 (Dupont Médical, Frouard, France). Both clinical and self-measurement of blood pressure are performed in this study.

* Clinical BP measurements are performed in the morning (from 8 am to noon), by doctors or nurses, in the patient's room or in the infirmary of the institute, after 10 minutes rest. All measurements are repeated three times, with intervals of 3 min on the left arm in a sitting position without replacing the cuff between the three measurements, according to the specific recommendations of the European Society of Hypertension.
* Self-measurements of BP are performed following the rule of 3 (3 measurements morning and evening during 3 consecutive days) according to the protocol proposed by the French society of hypertension. Self-measurements are performed by the subject her/himself in the room where he/she lives habitually. In case of difficulty, measurement are realized with the assistance of the nurse of the medical research team or of the institution.

Central blood pressure measurement Central BP values and aortic pressure waveform are obtained from the common carotid waveform using applanation tonometry. The PulsePen device (DiaTecne srl, Milan, Italy), a validated, easy to use, high-fidelity tonometer is used.

Pulse wave velocity PulsePen device is also used to measuring carotid-radial pulse wave velocity (PWV) which reflects upper limb arterial stiffness and carotid-femoral PWV corresponding to the aortic stiffness.

Follow-up data:

Medical research teams record every 3 months during a follow-up of 2 years deaths and following cardiovascular events: stroke, transient ischemic attack, myocardial infarction, unstable angina, acute pulmonary oedema, aortic aneurysm rupture, peripheral arterial thromboembolism, venous thrombosis and other major cardiovascular event. Moreover, a new assessment of autonomy, by ADL, and cognitive functions, by MMSE, are achieved in the cohort by the research teams one year and two year after the first visit.

ELIGIBILITY:
Inclusion Criteria:

* women and men aged 80 year old and over
* living in nursing home
* who signed the informed consent.

Exclusion Criteria:

* severe dementia (Mini Mental Status Examination: MMSE<12)
* a low level of autonomy (Activity of daily living: ADL≤2)
* under guardianship or "a measure of legal protection".

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This population-based study included 1200 voluntary subjects aged 80 and older, living in nursing home, included by four french university hospitals centre (Nancy, Dijon, Paris, Toulouse) and two Italian (Cesena, Verona).
Sampling Method: Non-Probability Sample
Enrollment: 1130 (Actual)
Dates: Start 2007-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Total Mortality | 2 years Follow-up

SECONDARY OUTCOMES:
Cardiovascular morbidity Cognitive decline | 2 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Athanase BENETOS, Professor, Principal Investigator — University Hospital of Nancy, department of geriatrics.
Locations (6):
- France (4):
  - University hospital of Dijon (Centre de Champmaillot), Dijon
  - Hôpital Broca, Paris
  - Hôpital La Grave, Toulouse
  - University hospital of Nancy, Vandœuvre-lès-Nancy
- Italy (2):
  - Hospital of Cesena, Cesena
  - Civil hospital Maggiore (Geriatrics), Verona

REFERENCES:
- [Background] Meaume S, Benetos A, Henry OF, Rudnichi A, Safar ME. Aortic pulse wave velocity predicts cardiovascular mortality in subjects >70 years of age. Arterioscler Thromb Vasc Biol. 2001 Dec;21(12):2046-50. doi: 10.1161/hq1201.100226. PMID 11742883
- [Background] Boshuizen HC, Izaks GJ, van Buuren S, Ligthart GJ. Blood pressure and mortality in elderly people aged 85 and older: community based study. BMJ. 1998 Jun 13;316(7147):1780-4. doi: 10.1136/bmj.316.7147.1780. PMID 9624064
- [Background] Satish S, Zhang DD, Goodwin JS. Clinical significance of falling blood pressure among older adults. J Clin Epidemiol. 2001 Sep;54(9):961-7. doi: 10.1016/s0895-4356(01)00360-2. PMID 11520657
- [Background] Askari M, Kiely DK, Lipsitz LA. Is pulse pressure a predictor of cardiovascular complications in a frail elderly nursing home population? Aging Clin Exp Res. 2004 Jun;16(3):206-11. doi: 10.1007/BF03327385. PMID 15462463
- [Background] Alecu C, Labat C, Kearney-Schwartz A, Fay R, Salvi P, Joly L, Lacolley P, Vespignani H, Benetos A. Reference values of aortic pulse wave velocity in the elderly. J Hypertens. 2008 Nov;26(11):2207-12. doi: 10.1097/HJH.0b013e32830e4932. PMID 18854762
- [Background] Benetos A, Adamopoulos C, Bureau JM, Temmar M, Labat C, Bean K, Thomas F, Pannier B, Asmar R, Zureik M, Safar M, Guize L. Determinants of accelerated progression of arterial stiffness in normotensive subjects and in treated hypertensive subjects over a 6-year period. Circulation. 2002 Mar 12;105(10):1202-7. doi: 10.1161/hc1002.105135. PMID 11889014
- [Background] Beckett NS, Peters R, Fletcher AE, Staessen JA, Liu L, Dumitrascu D, Stoyanovsky V, Antikainen RL, Nikitin Y, Anderson C, Belhani A, Forette F, Rajkumar C, Thijs L, Banya W, Bulpitt CJ; HYVET Study Group. Treatment of hypertension in patients 80 years of age or older. N Engl J Med. 2008 May 1;358(18):1887-98. doi: 10.1056/NEJMoa0801369. Epub 2008 Mar 31. PMID 18378519
- [Background] Salvi P, Lio G, Labat C, Ricci E, Pannier B, Benetos A. Validation of a new non-invasive portable tonometer for determining arterial pressure wave and pulse wave velocity: the PulsePen device. J Hypertens. 2004 Dec;22(12):2285-93. doi: 10.1097/00004872-200412000-00010. PMID 15614022
- [Derived] Salvi P, Grillo A, Gautier S, Labat C, Salvi L, Valbusa F, Baldi C, Rovina M, Simon G, Gao L, Tan I, Fabris B, Carretta R, Avolio AP, Parati G, Benetos A. Myocardial oxygen supply and demand imbalance predicts mortality in older nursing home residents: The PARTAGE study. J Am Geriatr Soc. 2024 Apr;72(4):1048-1059. doi: 10.1111/jgs.18752. Epub 2024 Jan 13. PMID 38217343
- [Derived] Mourad JJ, Agnoletti D, Labat C, Gautier S, Salvi P, Valbusa F, Hanon O, Toulza O, Manckoundia P, Fantin F, Rolland Y, Benetos A. Interest of Combined Blood Pressure Measurements in Very Old Frail Subjects: The PARTAGE Study. Am J Hypertens. 2018 Jul 16;31(8):950-956. doi: 10.1093/ajh/hpy077. PMID 30016415
- [Derived] Agnoletti D, Valbusa F, Labat C, Gautier S, Mourad JJ, Benetos A; PARTAGE study Investigators. Evidence for a Prognostic Role of Orthostatic Hypertension on Survival in a Very Old Institutionalized Population. Hypertension. 2016 Jan;67(1):191-6. doi: 10.1161/HYPERTENSIONAHA.115.06386. Epub 2015 Nov 23. PMID 26597824
- [Derived] Watfa G, Benetos A, Kearney-Schwartz A, Labat C, Gautier S, Hanon O, Salvi P, Joly L; PARTAGE study investigators. Do Arterial Hemodynamic Parameters Predict Cognitive Decline Over a Period of 2 Years in Individuals Older Than 80 Years Living in Nursing Homes? The PARTAGE Study. J Am Med Dir Assoc. 2015 Jul 1;16(7):598-602. doi: 10.1016/j.jamda.2015.01.098. Epub 2015 Mar 14. PMID 25783622
- [Derived] Miljkovic D, Perret-Guillaume C, Alla F, Salvi P, Erpelding ML, Benetos A. Correlation between peripheral blood pressure and pulse-wave velocity values in the institutionalized elderly persons 80 years of age and older: the PARTAGE study. Am J Hypertens. 2013 Feb;26(2):163-73. doi: 10.1093/ajh/hps042. Epub 2012 Dec 27. PMID 23382400
- [Derived] Benetos A, Gautier S, Labat C, Salvi P, Valbusa F, Marino F, Toulza O, Agnoletti D, Zamboni M, Dubail D, Manckoundia P, Rolland Y, Hanon O, Perret-Guillaume C, Lacolley P, Safar ME, Guillemin F. Mortality and cardiovascular events are best predicted by low central/peripheral pulse pressure amplification but not by high blood pressure levels in elderly nursing home subjects: the PARTAGE (Predictive Values of Blood Pressure and Arterial Stiffness in Institutionalized Very Aged Population) study. J Am Coll Cardiol. 2012 Oct 16;60(16):1503-11. doi: 10.1016/j.jacc.2012.04.055. Epub 2012 Sep 19. PMID 22999729
- [Derived] Valbusa F, Labat C, Salvi P, Vivian ME, Hanon O, Benetos A; PARTAGE investigators. Orthostatic hypotension in very old individuals living in nursing homes: the PARTAGE study. J Hypertens. 2012 Jan;30(1):53-60. doi: 10.1097/HJH.0b013e32834d3d73. PMID 22080223
- [Derived] Benetos A, Watfa G, Hanon O, Salvi P, Fantin F, Toulza O, Manckoundia P, Agnoletti D, Labat C, Gautier S; PARTAGE Study Investigators. Pulse wave velocity is associated with 1-year cognitive decline in the elderly older than 80 years: the PARTAGE study. J Am Med Dir Assoc. 2012 Mar;13(3):239-43. doi: 10.1016/j.jamda.2010.08.014. Epub 2010 Oct 20. PMID 21450208
- [Derived] Salvi P, Safar ME, Labat C, Borghi C, Lacolley P, Benetos A; PARTAGE Study Investigators. Heart disease and changes in pulse wave velocity and pulse pressure amplification in the elderly over 80 years: the PARTAGE Study. J Hypertens. 2010 Oct;28(10):2127-33. doi: 10.1097/HJH.0b013e32833c48de. PMID 20634719
- [Derived] Benetos A, Buatois S, Salvi P, Marino F, Toulza O, Dubail D, Manckoundia P, Valbusa F, Rolland Y, Hanon O, Gautier S, Miljkovic D, Guillemin F, Zamboni M, Labat C, Perret-Guillaume C. Blood pressure and pulse wave velocity values in the institutionalized elderly aged 80 and over: baseline of the PARTAGE study. J Hypertens. 2010 Jan;28(1):41-50. doi: 10.1097/HJH.0b013e328332b879. PMID 19809365